CLINICAL TRIAL: NCT00091052
Title: Contrast-Enhanced Radiotherapy With GM-CSF Immune Stimulation - Phase I/II Clinical Center Treatment Trial
Brief Title: Radiation Therapy and Sargramostim in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sirius Medicine (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000383147; SIRIUS-1053285; SIRIUS-01
Record Dates: First submitted 2004-09-07; First posted 2004-09-08 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2006-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — sargramostim; Radiotherapy

INTERVENTIONS:
Biological: sargramostim
Radiation: radiation therapy

SUMMARY:
RATIONALE: Colony-stimulating factors such as sargramostim increase the number of immune cells found in bone marrow or peripheral blood. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining radiation therapy with sargramostim may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects of giving radiation therapy together with sargramostim and to see how well it works in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of contrast-enhanced high-dose radiotherapy administered with sargramostim (GM-CSF) in patients with advanced solid malignancies.
* Determine immune response in patients treated with this regimen.
* Determine tumor response in patients treated with this regimen.

OUTLINE: Patients are stratified according to prior therapy (biopsy or simple surgery vs radical surgery, chemotherapy, or radiotherapy).

Patients receive a contrast agent intratumorally followed by a single fraction of kilovoltage radiotherapy. Beginning 24 hours after radiotherapy, patients receive sargramostim (GM-CSF) intratumorally continuously for 1 week and then subcutaneously for 2 weeks. Patients with lung tumors receive GM-CSF by inhalation twice daily for 1 week and then every other week for a total of 3 weeks of drug treatment.

Treatment may repeat in several weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 8 weeks.

PROJECTED ACCRUAL: A total of 47 patients (12 for phase I and 35 for phase II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid malignancy

  * Advanced disease
* Radiotherapy is appropriate treatment (i.e., radio-responsive)

  * No tumors beyond the reach of kilovoltage beam (e.g., > 15 cm beneath the skin)
* At least 1 lesion accessible to needle localization and catheter placement
* May be refractory to prior chemotherapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* 0-4

Life expectancy

* At least 2 months

Hematopoietic

* Hemoglobin ≥ 10 g/dL (RBC transfusion allowed)
* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3 (transfusion independent)
* No excessive leukemic blasts
* No bleeding diathesis

Hepatic

* PT and PTT ≤ 1.5 times upper limit of normal (ULN)
* AST or ALT < 2 times ULN
* Alkaline phosphatase < 2 times ULN

Renal

* Creatinine < 1.5 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* No contraindication to MRI or CT scan
* No medical or psychiatric condition that would preclude giving informed consent
* Able to lie flat for 1 hour
* No known hypersensitivity to sargramostim (GM-CSF) or any of its components

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior biologic therapy allowed
* No concurrent biologic therapy

Chemotherapy

* See Disease Characteristics
* No concurrent chemotherapy

Endocrine therapy

* Concurrent hormonal therapy allowed

Radiotherapy

* Prior radiotherapy to planned treatment site allowed
* No other concurrent radiotherapy to planned treatment site

Surgery

* Prior surgery allowed

Other

* More than 14 days since prior radiosensitizers
* No other concurrent investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-07; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Toxicity as measured by the Southwest Oncology Group Performance Status and Toxicity Criteria on day 1 and in weeks 4, 12, and 20

SECONDARY OUTCOMES:
Immune and tumor response as measured by reverse transcriptase polymerase chain reaction (RT-PCR) and CT scan on day 1 and in weeks 2, 3, 4, 12, and 20 or weeks 4, 12, and 20

CONTACTS AND LOCATIONS:
Overall Officials: Michael D. Weil, MD, Study Chair — Sirius Medicine
Locations (1):
- Sirius Medicine, LLC, Loveland, Colorado, United States